CLINICAL TRIAL: NCT02237365
Title: A Pilot Phase II Randomized Controlled Double Blind Trial of 81mg Aspirin Daily vs. 1000 mg Aspirin Daily vs. Placebo as Adjunctive Therapy in HIV Negative Adults With Tuberculous Meningitis
Brief Title: A Pilot Study of Adjunctive Aspirin for the Treatment of HIV Negative Adults With Tuberculous Meningitis
Acronym: AspirinTBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23TB
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Tuberculous Meningitis
Keywords: neurological disability; tuberculous meningitis (TBM); safety; aspirin; efficacy
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 81mg aspirin (Experimental): Aspirin 81mg daily for 60 days
  Interventions: Drug: 81mg aspirin
- 1000mg aspirin (Experimental): Aspirin 1000mg daily for 60 days
  Interventions: Drug: 1000mg aspirin
- Placebo (Placebo Comparator): Visually matched placebo daily for 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 81mg aspirin — 1 tablet of 81mg aspirin and 2 tablets of placebo (visually matched to 500mg aspirin) daily for 60 days
  Arms: 81mg aspirin
Drug: 1000mg aspirin — 1 tablet of 81mg placebo (visually matched to 81mg aspirin) and 2 tablets of 500mg aspirin daily for 60 days
  Arms: 1000mg aspirin
Drug: Placebo — 1 tablet of 81mg placebo (visually matched to 81mg aspirin) and 2 tablets of 500mg placebo (visually matched to 500mg aspirin) daily for 60 days
  Arms: Placebo

SUMMARY:
Tuberculous meningitis is a severe brain infection which often causes disability and death even when treated with the best available treatment. Aspirin is a type of anti-inflammation drug which can reduce the inflammatory response in brains of patients with tuberculous meningitis, and therefore may decrease some of the most severe outcomes. This study compares the use of aspirin (at 2 different doses) versus placebo as an additional therapy to the standard treatment to see if aspirin is safe and helpful in reducing disability and death from tuberculous meningitis. Patients will be treated with aspirin or placebo for 60 days and followed up while on standard treatment for 8 months.

DETAILED DESCRIPTION:
The study is a parallel group, double blind, randomised, placebo controlled trial of 60 days treatment with placebo vs. 81mg daily dose vs. 1000mg daily dose aspirin for the treatment of HIV-uninfected adults with tuberculous meningitis.

All patients will receive standard anti-tuberculous chemotherapy and adjunctive dexamethasone, according to Viet Nam National Tuberculosis Programme guidelines. Participants will be stratified by Medical Research Council UK disease severity grade, and randomized at enrollment to one of three study arms (1:1:1 ratio). Patients will be admitted to hospital for at least the first 14 days of study treatment enabling real-time active surveillance of any adverse events after which they will be discharged according to clinical care with continued monitoring.

A schedule of clinical and laboratory monitoring including lumbar puncture, pharmacokinetic assessment of peripheral blood monocyte/macrophage antimicrobial activity, clinical assessments, brain magnetic resonance imaging (MRI) and neurological assessment will manage patient safety and capture study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or above.
* Suspected TBM and anti-tuberculosis chemotherapy either planned or started
* Less than 3 days of anti-tuberculosis chemotherapy taken for the current infection
* Patient or representative (if the patient is unable) is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* HIV infection (negative rapid test or Elisa test is required)
* Unlikely, for any reason, to be able to have an MRI brain scan within 5 days (120 hours) of randomisation
* Known or suspected infection with multi-drug resistant tuberculosis (resistant to at least isoniazid and rifampicin)
* Unable to take isoniazid, rifampicin, or pyrazinamide at recommended doses for any reason
* History of diagnosed peptic ulceration or gastro-intestinal bleeding
* Active gastro-intestinal bleeding is suspected
* Taken >1 dose of aspirin (at any dose) or any other non-steroidal anti-inflammatory drugs for any reason within 2 weeks of screening
* Aspirin considered mandatory for any reason by the attending physician
* Aspirin considered to be contraindicated for any reason by the attending physician
* Pregnancy or breast feeding (negative urine pregnancy test for all females of child-bearing age)
* Dexamethasone considered to be contraindicated for any reason by the attending physician
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Number of episodes of either cerebral bleeding or clinically significant upper-gastro-intestinal bleeding (composite endpoint) | 60 days
  Primary Safety Endpoint: Number of episodes of:
  1. Cerebral bleeding confirmed by brain imaging and/or
  2. Clinically significant upper-gastro-intestinal bleeding, defined as: a) Vomiting fresh or changed blood of any volume; b) Melena; c) Unexplained drop in haemoglobin concentration of >2g/L or; d) Greater than 5mls of fresh or changed blood aspirated from nasogastric tube
Number of episodes of MRI-proven brain infarction or death (composite endpoint) | 60 days
  Primary Efficacy Endpoint: Number of episodes of
  1. MRI-proven brain infarction and/or
  2. Death

SECONDARY OUTCOMES:
Time to death | 240 days
Number of grade 3&4 and serious adverse events | 60 days
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) definitions
Duration of hospital stay | 240 days
  Number of days admitted to hospital during the study period
Neurological disability score | 60 days
  Assessed by the modified Rankin score and Glasgow outcome score
Neurological disability score | 240 days
  Assessed by the modified Rankin score and Glasgow outcome score
Resolution of cerebrospinal fluid (CSF) inflammation | 30 days
  Evaluated by measurement of CSF leucocytes, protein, glucose, cytokines (TNF-α, IL-1β, IL-8, IL-10, IFNγ) and eicosanoids (15-epi-Lipoxin, Lipoxin A4, LTB4, PGE2, TBXB2, PGD2)
Antimicrobial activity of peripheral blood monocyte/macrophages | 240 days
  Difference between measured antimicrobial activity at baseline and 240 days
Proportion of patients with MRI-proven brain infarction | 240 days

CONTACTS AND LOCATIONS:
Overall Officials: Guy Thwaites, MD, PhD, Principal Investigator — Oxford University of Clinical Research; Nguyen H Phu, MD, PhD, Principal Investigator — Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Mai NTH, Dobbs N, Phu NH, Colas RA, Thao LTP, Thuong NTT, Nghia HDT, Hanh NHH, Hang NT, Heemskerk AD, Day JN, Ly L, Thu DDA, Merson L, Kestelyn E, Wolbers M, Geskus R, Summers D, Chau NVV, Dalli J, Thwaites GE. A randomised double blind placebo controlled phase 2 trial of adjunctive aspirin for tuberculous meningitis in HIV-uninfected adults. Elife. 2018 Feb 27;7:e33478. doi: 10.7554/eLife.33478. PMID 29482717
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org